CLINICAL TRIAL: NCT07007156
Title: Is a Positive NECPAL in ICU Patients Associated With Higher Mortality
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-74
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Disease
Keywords: Acute Disease; Intensive Care Unit
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NECPAL positive — This group has a positive result for NECPAL scale

SUMMARY:
The aim of the present study is to evaluate the usefulness of the NECPAL scale in identifying Intensive Care Unit (ICU)-admitted patients at higher risk of dying within 90 days of ICU admission

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following inclusion criteria may be included in the study:
* Men and women aged 75 years or older.
* Admission to the ICU of the study center.
* Legal capacity to provide informed consent.
* Signed informed consent for study inclusion, either by the participant or their legal representative.

Exclusion Criteria:

Participants who meet any of the following exclusion criteria may not be included in the study:

-Death within the first 24 hours of ICU admission.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 years or older who are admitted to an ICU
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | From baseline to 90-day
  Patients who dye at 90-day from ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gutiérrez, MD, Principal Investigator — CSAPG
Locations (1):
- CSAPG, Sant Pere de Ribes, Barcelona, Spain